CLINICAL TRIAL: NCT02976493
Title: Elotuzumab Safety Surveillance In Japanese Patients With Relapse Or Refractory Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-179
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MM patients receiving elotuzumab: Non-Interventional Study of all patients with relapsed or refractory multiple myeloma (MM) who are beginning to receive elotuzumab at the selected sites.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
BMS will conduct a regulatory postmarketing surveillance (PMS) to evaluate the safety of elotuzumab in clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All patients with relapsed or refractory multiple myeloma who are beginning to receive elotuzumab at the selected sites will be included in this surveillance study

Exclusion Criteria:

* Not Applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed or refractory multiple myeloma who are beginning to receive elotuzumab at healthcare facilities in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events(AE) to elotuzumab in real-world practice in Japan | Up to 72 weeks
Incidence of immune-related (IR) adverse events to elotuzumab in real-world practice in Japan | Up to 72 weeks
  immune-related (IR) adverse events are defined as: 1) AEs that are related to elotuzumab per investigator and 2) are consistent with an inflammatory process.
Number of patients who achieve a Stringent complete response (sCR) as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks
Number of patients who achieve a Complete response (CR) as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks
Number of patients who achieve a Very good partial response (VGPR) as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks
Number of patients who achieve a Partial response (PR) as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks
Number of patients who achieve a Progressive Disease (PD) as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks
Number of patients who achieve a Relapse from complete response as measured by International Myeloma Working Group (IMWG) criteria | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx